CLINICAL TRIAL: NCT02946060
Title: The Music Activity INTervention for Adherence Improvement Through Neurological Entrainment - II
Acronym: MAINTAIN-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dr. David Alter, Principal Investigator, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-9839
Record Dates: First submitted 2016-09-19; First posted 2016-10-26 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Sound Recordings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (Sham Comparator): Participants in this intervention will receive the minimal standard of care provided at the Cardiac Rehabilitation and Prevention Program at Toronto Rehabilitation Institute. Participants will receive an iPod with a silent track or white noise.
  Interventions: Other: Usual Care
- Audiobooks (Active Comparator): Participants in this arm will receive iPods with Audiobooks based on their preferred genres.
  Interventions: Other: Audiobooks
- Tempo-pace Synchronized Playlists (Experimental): Participants in this arm will receive audio playlists synchronized to their exercise pace. Rhythmic enhancements will be added to the playlists during either month 2 or month 3 of the study.
  Interventions: Other: Tempo-pace synchronized playlists

INTERVENTIONS:
Other: Audiobooks — iPods with audiobooks
  Arms: Audiobooks
Other: Tempo-pace synchronized playlists — Playlists with or without RAS
  Arms: Tempo-pace Synchronized Playlists
Other: Usual Care — iPods containing either a silent track or white noise
  Arms: Usual Care

SUMMARY:
This study (MAINTAIN -II) aims to examine the effect of audio playlists [with or without Rhythmic Auditory Stimulation (RAS)] on the weekly volume of physical activity. Participants will be randomized into 3 Interventions: Control (standard, usual care), Audiobook, or Tempo-pace Synchronized Playlists (TSP). The investigators also aim to explore the effects of these interventions on mood, perceived exertion and dissociative attention among patients participating in cardiac rehabilitation.

DETAILED DESCRIPTION:
Physical activity is associated with a 35% decrease in cardiovascular mortality - a direct result of exercise on the vasculature and an indirect result of exercise lowering CVD risk factors such as lipids and blood pressure. With physical inactivity being one of the major independent risk factors for CVD, structured exercise cardiac rehabilitation programs have been implemented to encourage adherence to physical activity among patients with cardiac related issues. Clinical trial evidence has demonstrated irrefutable mortality and morbidity benefits associated with cardiac rehabilitation especially among patients with established CVD. The mechanisms for improved outcomes are likely multifactorial, including improved preventative self-management, physical activity volume, and cardiopulmonary fitness. Unfortunately the real-world outcome benefits associated with cardiac rehabilitation are undermined by behavioural attrition, with programmatic drop out and suboptimal physical activity adherence patterns that mirror the broader healthy population who are not enrolled in cardiac rehabilitation.

Unfortunately the real-world outcome benefits associated with cardiac rehabilitation are undermined by attrition rates of up to 50% post rehabilitation. The goal would therefore be to introduce a co-intervention that encourages long-term exercise adherence for maximal health improvements in cardiac rehabilitation populations, which might also have broader applicability to other non-cardiac rehab populations.

The prior study, The Music Activity INTervention for Adherence Improvement through Neurological entrainment (MAINTAIN -1), examined the use of Tempo Synchronized Playlists (TSP) on improving exercise adherence within the cardiac rehabilitation program. Weekly volumes of physical activity were compared between groups assigned to 3 interventions: control group receiving Usual Care, TSP, and Tempo-pace Synchronized Playlists with Rhythmic Auditory Stimulation (RAS). Rhythmic Auditory Stimulation is a neurological rehabilitation technique used to accentuate tempo-pace synchrony. The group assigned to the TSP intervention demonstrated a significantly higher volume in weekly exercise than the usual care control group. Furthermore, the group randomized to TSP with RAS partook in twice the amount of weekly physical activity than the TSP group without RAS. Our prior study had several limitations including small sample size and an inability to examine the mechanisms by which RAS tempo-based audio-playlist synchronization mediated increases in physical activity.

The objective of this current study is to build on our previous research by examining the reproducibility of efficacy and exploring the mechanisms such as mood, perceived exertion and dissociative attention, by which the preference-based tempo-pace synchronized playlists improve exercise adherence among patients participating in cardiac rehabilitation. Participants will be randomized into 3 Interventions: Usual Care, Audiobooks, and TSP, that will be assigned during months 2 and 3 of the program. The Usual Care group will feature a nested design by which half patients will randomized to receive a silent track during month 2, and the other half will receive white noise. This sequence will be reversed during month 3. Within the TSP intervention, 2 nested designs will be tested. The first will test RAS with non-RAS. Half of the patients will be randomized to receive TSP with RAS during month 2 of the study, while the other half will receive TSP without RAS during month 2. The sequence will be reversed in month 3. The second will determine the effect on training by comparing 'active' vs. 'passive'. Within the active group, participants will be trained on how to exercise with the music. The passive group will not be trained.

Cardiac Rehabilitation provides an ideal test-case program by which to examine music co-interventions, as it mirrors the behavioural attrition experienced in other structured or unstructured exercise activities. Additionally, a music tempo-pace synchronization strategy is appropriate in such a setting as it helps to regulate the exercise pace prescribed to each patient by the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known cardiovascular disease who are participating in and have been declared medically stable for outpatient cardiac rehabilitation
* Patients must be at least 18 years of age
* Patients must have received at least one exercise prescription that includes consistent walking and/or running (no high interval training or stationary machines)

Exclusion Criteria:

* Participants unable to wear the iPod device or activity monitoring device due to medical or non-medical issues
* Participants with significant communication impairments
* Participants currently enrolled in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Average volume of physical activity per week per intervention | 12 weeks
  The activity monitor will be worn each week for 12 weeks. Average minutes of physical activity per week will be compared between groups.

SECONDARY OUTCOMES:
Affect measured by Feeling Scale | Biweekly for the duration of 12 weeks
  During participant's biweekly exercise session, scores on the Feeling Scale will be recorded per lap.
Arousal measured by Score on Felt Arousal | Biweekly for the duration of 12 weeks
  During participants biweekly exercise session, scores on the Felt Arousal Scale will be recorded per lap
Perceived Exertion measured by Rate of Perceived Exertion Scale | Biweekly for the duration of 12 weeks
  During participants biweekly exercise session, scores on the Rate of Perceived Exertion Scale (RPE) will be recorded per lap.
Dissociative Attention measured by the Tammen's Scale | Biweekly for the duration of 12 weeks
  During participants biweekly exercise session, scores on the Tammen's scale will be recorded per lap.
Focus measured by the Focus Questionnaire | Biweekly for the duration of 12 weeks
  During participants' biweekly exercise session, focus on the audio in the headphones will be recorded at the end of the exercise.
Pacing of Exercise | Biweekly for the duration of 12 weeks
  Number of steps in one minute will be counted during exercise session.
Lap time | Biweekly for the duration of 12 weeks
  Time taken to complete one lap will be recorded for each biweekly exercise session.
Playcounts | 8 week duration
  Number of plays of the audio file per week will be recorded
Future Hospitalizations and/or Mortality | Within 2 years
  Participants will be tracked longitudinally throughout health service encounters including physician visits, hospitalizations, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Alter, MD,PhD,FRCPC, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Cardiac Rehabilitation and Prevention Program, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alter DA, Wijeysundera HC, Franklin B, Austin PC, Chong A, Oh PI, Tu JV, Stukel TA. Obesity, lifestyle risk-factors, and health service outcomes among healthy middle-aged adults in Canada. BMC Health Serv Res. 2012 Aug 4;12:238. doi: 10.1186/1472-6963-12-238. PMID 22863333
- [Background] Alter DA, Zagorski B, Marzolini S, Forhan M, Oh PI. On-site programmatic attendance to cardiac rehabilitation and the healthy-adherer effect. Eur J Prev Cardiol. 2015 Oct;22(10):1232-46. doi: 10.1177/2047487314544084. Epub 2014 Jul 30. PMID 25079239
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Brewer, BW., Van Raalte, JL, & Linder, DE. (1996). Attentional Focus and Endurance Performance. Applied Research in Coaching and Athletics Annual. 11:1-14.
- [Background] Brownley KA, McMurray RG, Hackney AC. Effects of music on physiological and affective responses to graded treadmill exercise in trained and untrained runners. Int J Psychophysiol. 1995 Apr;19(3):193-201. doi: 10.1016/0167-8760(95)00007-f. PMID 7558986
- [Background] Chen JL, Zatorre RJ, Penhune VB. Interactions between auditory and dorsal premotor cortex during synchronization to musical rhythms. Neuroimage. 2006 Oct 1;32(4):1771-81. doi: 10.1016/j.neuroimage.2006.04.207. Epub 2006 Jun 14. PMID 16777432
- [Background] Davies P, Taylor F, Beswick A, Wise F, Moxham T, Rees K, Ebrahim S. Promoting patient uptake and adherence in cardiac rehabilitation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007131. doi: 10.1002/14651858.CD007131.pub2. PMID 20614453
- [Background] Goel K, Lennon RJ, Tilbury RT, Squires RW, Thomas RJ. Impact of cardiac rehabilitation on mortality and cardiovascular events after percutaneous coronary intervention in the community. Circulation. 2011 May 31;123(21):2344-52. doi: 10.1161/CIRCULATIONAHA.110.983536. Epub 2011 May 16. PMID 21576654
- [Background] Hardy, CJ., & Rejeski, WJ. (1989). Not What, but How One Feels: the Measurement of Affect During Exercise. J. Sport Exerc Psychol. 11:304-317
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Kendzierski D, DeCarlo KJ. Physical Activity Enjoyment Scale: Two validation studies. Journal of Sport & Exercise Psychology. 1991;13(1):50-64.
- [Background] Measuring Enjoyment of Physical Activity in Children: Validation of the Physical Activity Enjoyment Scale. J Appl Sport Psychol. 2009 Jan 1;21(S1):S116-S129. doi: 10.1080/10413200802593612. PMID 20209028
- [Background] Nakamura PM, Pereira G, Papini CB, Nakamura FY, Kokubun E. Effects of preferred and nonpreferred music on continuous cycling exercise performance. Percept Mot Skills. 2010 Feb;110(1):257-64. doi: 10.2466/PMS.110.1.257-264. PMID 20391890
- [Background] Nocon M, Hiemann T, Muller-Riemenschneider F, Thalau F, Roll S, Willich SN. Association of physical activity with all-cause and cardiovascular mortality: a systematic review and meta-analysis. Eur J Cardiovasc Prev Rehabil. 2008 Jun;15(3):239-46. doi: 10.1097/HJR.0b013e3282f55e09. PMID 18525377
- [Background] Pinch, TJ., & Bijsterveld, K. (2012). The Oxford Handbook of Sound Studies. New York: Oxford University Press.
- [Background] Simpson SD, Karageorghis CI. The effects of synchronous music on 400-m sprint performance. J Sports Sci. 2006 Oct;24(10):1095-102. doi: 10.1080/02640410500432789. PMID 17115524
- [Background] Svebak, S., & Murgatroyd, S. (1985). Metamotivational dominance: A multi-method validation of reversal theory constructs. Journal of Personality and Social Psychology. 48: 107-116.
- [Background] Tammen, VV. (1996). Elite middle and long distance runner's associative/dissociative coping. J. Apple. Sport Psychol. 8:1-810
- [Background] Taylor RS, Unal B, Critchley JA, Capewell S. Mortality reductions in patients receiving exercise-based cardiac rehabilitation: how much can be attributed to cardiovascular risk factor improvements? Eur J Cardiovasc Prev Rehabil. 2006 Jun;13(3):369-74. doi: 10.1097/01.hjr.0000199492.00967.11. PMID 16926666
- [Background] Thompson DR, Bowman GS, Kitson AL, de Bono DP, Hopkins A. Cardiac rehabilitation services in England and Wales: a national survey. Int J Cardiol. 1997 May 23;59(3):299-304. doi: 10.1016/s0167-5273(97)02951-3. PMID 9183047
- [Background] Turk-Adawi KI, Oldridge NB, Tarima SS, Stason WB, Shepard DS. Cardiac rehabilitation patient and organizational factors: what keeps patients in programs? J Am Heart Assoc. 2013 Oct 21;2(5):e000418. doi: 10.1161/JAHA.113.000418. PMID 24145743
- [Background] WHO. Preventing chronic diseases: A vital investment (2005) [accessed September 20, 2015].http://www .who.int/chp /chronic_disease_report/full_report .pdf.
- [Background] Woodcock J, Franco OH, Orsini N, Roberts I. Non-vigorous physical activity and all-cause mortality: systematic review and meta-analysis of cohort studies. Int J Epidemiol. 2011 Feb;40(1):121-38. doi: 10.1093/ije/dyq104. Epub 2010 Jul 14. PMID 20630992